CLINICAL TRIAL: NCT04917913
Title: Efficacy of a Digestive Enzyme Blend: A Randomized, Double-Blind, Placebo-controlled Trial
Brief Title: Efficacy of a Digestive Enzyme Blend
Acronym: MULO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Deerland Enzymes (Industry)
Collaborators: Kennesaw State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: Digestive Enzymes
Record Dates: First submitted 2021-05-26; First posted 2021-06-08 (Actual); Last update posted 2021-06-08 (Actual); Status verified 2021-06

CONDITIONS: Digestive Health; Indigestion; Protein Digestion; Carbohydrate Digestion; Fat Digestion; Satiety
MeSH Terms: conditions — Dyspepsia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Subjects will be administered 3 daily doses (one per meal) of digestive enzymes (50mg), in a capsule, for 30 days
  Interventions: Dietary Supplement: Digestive enzyme blend
- Placebo (Placebo Comparator): Subjects will be administered 3 daily doses (one per meal) of digestive enzymes (50mg), in a capsule, for 30 days
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Digestive enzyme blend — Subjects will take 3 capsules (one per meal) of digestive enzymes (50mg) daily for 30 days.
  Arms: Intervention
Dietary Supplement: Placebo — Subjects will take 3 capsules (one per meal) of a placebo (50mg) daily for 30 days.
  Arms: Placebo

SUMMARY:
The purpose of this study is to investigate the effect of a digestive enzyme supplement (three times per day for 30 days) on gastrointestinal distress (GID) and body composition (body mass and body fat percentage) in healthy men and women (18 - 55 years of age) who experience regular GID (3 - 6 episodes of GID per month).

DETAILED DESCRIPTION:
Pre-Screening: Subjects will first undergo a pre-screening visit with the PI. The PI will go over the COVID-19 screening as well as the study screening for inclusion and exclusion criteria. Subjects will be given information regarding the study details, location of the study, and parking during this pre-screening visit as well.

Visit 1: This session will take place at the Exercise Physiology Laboratory (Prillaman 1102 - Kennesaw State University) and subjects will be asked to arrive fasted (8-10 hours). Subjects will be informed of the purpose, risks, and benefits of the study. They will be asked to review and sign this consent form. Subjects may ask questions at any time. They will then complete a Health History Questionnaire (HHQ) consisting of medical, physical activity, diet, and supplementation history. Following completion of this consent and the HHQ a member of the research team will take subjects to assess height, weight, and body composition (assessments described below). Immediately following the body composition assessment, they will be asked to fill out a series of questionnaires. These questionnaires will be electronic and will require subjects to use a computer as well as applications on their phone (surveys and applications described below).

A member of the research team will describe how to use the applications and computer programs: 1) Cronometer (for dietary tracking); 2) MyGiHealth (for GID tracking); and 3) SurveyMonkey (for GID tracking and supplement compliance tracking). Once subjects have completed all surveys a member of the research team will then distribute their first 30 day allotment of supplement (blinded, randomly assigned enzyme or placebo - both are 200 mg per pill) and provide subjects with instructions on how to take the supplement (3 times per day - right before a meal - for example right before breakfast, lunch, and dinner). They will then be informed on how to track their GID and diet throughout the 30 days of supplementation (described below). Lastly, subjects will be given their return date for Visit 2 and work with the research team member on a time that works for them.

Visit 2: Subjects will return to the lab for Visit 2 following 30 days of supplementation. During visit 2, they will have their body composition reassessed, as well as complete all GID surveys as they did during Visit 1. Further, a member of the research team will ensure that they completed all proper tracking of diet and GID during the 30 day supplementation period. Subjects will then work with the research team member to determine a Visit 3 date. Visit 3 will be at least 7 days after Visit 2.

Visit 3 and Visit 4: Visits 3 and 4 will be similar to Visits 1 and 2, respectively. However, subjects will not complete the informed consent form again and will not have to download/install the applications, as they will have completed this during Visit 1. During Visits 3 and 4, they will first have their body composition reassessed and fill out questionnaires (GID) (same as Visit 1 and 2). Further, subjects will be asked to take the supplement they did not receive during the first 30 days, for 30 days following Visit 3 (still blind to both the participants and research team). Subjects again will be asked to track their diet and GID during the 30 days of supplementation between Visits 3 and 4 (see tracking below). Following completion of Visit 4, subjects will receive their body composition results from visits 4.

ELIGIBILITY:
Inclusion Criteria:

* Be 18 - 55 years of age.
* Experience occasional gastrointestinal distress - 3 -6 episodes per month.
* Gastrointestinal distress may be defined as constipation, upset stomach, diarrhea, stomach cramping, bowel incontinence, heart-burn, acid reflux, gastroesophageal reflux, bloating or swelling of the belly, nausea or vomiting

Exclusion Criteria:

* Currently taking prescription medications for gastrointestinal distress.
* Taking prescription medications that may be impacted by enzyme consumption.
* Taking steroidal medications.
* Currently ill. Have a diagnosed severe gastrointestinal disorder including: fissures, abscesses, or hemorrhoids.
* Have a greater than 30 kg/m2 BMI.
* Currently pregnant or attempting to get pregnant.
* Do not have access to a cell phone or computer daily.
* Are being treated by a clinician for GI disease.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-05-10 (Actual); Primary Completion 2022-01-31 (Estimated); Study Completion 2022-01-31 (Estimated)

PRIMARY OUTCOMES:
Gastrointestinal Distress | 30 days
  Analyze change in gastrointestinal distress symptoms obtained from questionnaires from baseline to 30 days.

CONTACTS AND LOCATIONS:
Overall Officials: Trisha VanDusseldorp, PhD, Principal Investigator — Kennesaw State University
Locations (1):
- Kennesaw State University, Kennesaw, Georgia, United States

IPD SHARING:
Plan to Share IPD: No